CLINICAL TRIAL: NCT03222570
Title: An Adaptive Algorithm-Based Approach to Treatment for Adolescent Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PSYCH-2017-25767; R01MH113748 (NIH)
Record Dates: First submitted 2017-07-13; First posted 2017-07-19 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Interpersonal Psychotherapy; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IPT-A Adaptive Treatment Strategy (Experimental): Adolescents begin with an initial treatment plan of 12 weekly sessions of interpersonal psychotherapy for depressed adolescents (IPT-A). Depressive symptoms will be assessed at week 4 and week 8 of therapy. If an adolescent demonstrates an insufficient response at either time point, the adolescent will be randomized a second time to either an increased dose of IPT-A (sessions scheduled twice per week for 4 weeks;16 sessions total) or the addition of a selective serotonin reuptake inhibitor (SSRI).
  Interventions: Behavioral: Interpersonal Psychotherapy for Depressed Adolescents; Drug: Selective Serotonin Reuptake Inhibitor
- Usual Care (Active Comparator): Therapists will implement therapy procedures that they usually use and believe to be effective in clinical practice. Therapists will use whatever methods they usually use to make decisions regarding the frequency of therapy sessions and whether to refer the adolescent to start an SSRI.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Depressed Adolescents — IPT-A is an evidence-based intervention that aims to decrease depressive symptoms by helping adolescents improve their relationships and interpersonal interactions. It addresses one or more of four interpersonal problem areas: grief, role disputes, role transitions, and interpersonal deficits. The primary treatment techniques in IPT-A include emotion identification/expression, linking interpersonal events to mood, communication analysis, communication skill building, decision analysis, role playing, and assignment of interpersonal experiments (i.e. homework). In clinical trials, depressed adolescents treated with IPT-A demonstrated fewer depressive symptoms and better psychosocial functioning post-treatment than adolescents in control conditions.
  Arms: IPT-A Adaptive Treatment Strategy
Drug: Selective Serotonin Reuptake Inhibitor — Fluoxetine, escitalopram, citalopram, fluvoxamine, or sertraline
  Arms: IPT-A Adaptive Treatment Strategy
Other: Usual Care — Therapists will implement therapy procedures that they usually use and believe to be effective in clinical practice. Therapists will use whatever methods they usually use to make decisions regarding the frequency of therapy sessions and whether to refer the adolescent to start an SSRI
  Arms: Usual Care

SUMMARY:
The purpose of this study is to evaluate the effectiveness of two adaptive treatment strategies (ATSs) for adolescent depression. The ATSs include delivery of an evidence-based psychotherapy (interpersonal psychotherapy for depressed adolescents, IPT-A), systematic symptom monitoring, and an empirically-derived algorithm that specifies whether, when, and how to augment IPT-A. Two hundred depressed adolescents (age 12-18) will be recruited to participate in a 16-week sequential multiple assignment randomized trial conducted in outpatient community mental health clinics. Adolescents will be randomized to the IPT-A ATS condition or the community clinic's usual care (UC). Adolescents in the IPT-A ATS condition who are insufficient responders will be randomized a second time to the addition of a selective serotonin reuptake inhibitor (SSRI) or more intensive IPT-A (delivered twice per week). Research assessments will be administered at baseline and at weeks 4, 8, 12, 16, and 36.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-V criteria for a primary diagnosis of Major Depressive Disorder, Persistent Depressive Disorder, or Depressive Disorder NEC
* Current significant depressive symptoms (based on Children's Depression Rating Scale - Revised [CDRS-R])
* Current impairment in psychosocial functioning (based on Children's Global Assessment Scale [CGAS])

Exclusion Criteria:

* Non English-speaking
* Meet DSM-V criteria for bipolar disorder, psychosis, anorexia nervosa, substance use disorder, autism spectrum disorder, or intellectual disability disorder.
* Adolescents who are actively suicidal with a plan and/or intent who are assessed to need a higher level of care than outpatient treatment due to safety risk will be referred for appropriate level of stabilization. Once stabilized, the adolescent can be re-evaluated for eligibility to participate in the study.
* Currently taking medication for a psychiatric diagnosis other than ADHD

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
All data resulting from the proposed project will be shared via the National Database for Clinical Trials (NDCT).
Supporting Information: Study Protocol

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IPT-A Adaptive Treatment Strategy | Usual Care
Started | 57 | 33
Completed | 40 | 27
Not Completed | 17 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IPT-A Adaptive Treatment Strategy | Usual Care | Total
Number analyzed (Participants) | 57 | 33 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 57 | 33 | 90
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (1.6) | 14.2 (2.0) | 14.6 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 21 | 62
  Male | 16 | 12 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 46 | 24 | 70
  Unknown or Not Reported | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 43 | 24 | 67
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 57 | 33 | 90

OUTCOME MEASURES:

1. Primary Outcome: Children's Depression Rating Scale - Revised
Description: Minimum value: 17 Maximum value: 113 Higher scores indicate worse outcome
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-A Adaptive Treatment Strategy | Usual Care
Number analyzed (Participants) | 57 | 33
score on a scale | 36.0 (11.3) | 37.5 (11.7)
Statistical Analysis 1: Comparison: IPT-A Adaptive Treatment Strategy vs Usual Care; Test type: Superiority; p = 0.76, Regression, Linear; Estimated mean difference = -0.88, 95% CI 2-sided [-6.56 to 4.7] — Mean difference estimated from fitting a linear regression model adjusting for baseline value of the measure

2. Secondary Outcome: Children's Global Assessment Scale
Description: Measure of general psychosocial functioning Minimum score: 1 Maximum score: 100 A higher score indicates a better outcome
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-A Adaptive Treatment Strategy | Usual Care
Number analyzed (Participants) | 57 | 33
score on a scale | 61.8 (9.5) | 63.3 (12.1)
Statistical Analysis 1: Comparison: IPT-A Adaptive Treatment Strategy vs Usual Care; Test type: Superiority; p = 0.32, Regression, Linear; Estimated mean difference = -2.52, 95% CI 2-sided [-7.42 to 2.3] — Mean difference estimated from fitting a linear regression model adjusting for baseline value of the measure

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | IPT-A Adaptive Treatment Strategy | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/33
Other Adverse Events (participants affected / at risk) | 10/57 | 5/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPT-A Adaptive Treatment Strategy (N=57) | Usual Care (N=33)
Emergent or worsening suicidal ideation (Psychiatric disorders) | 10 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT03222570/Prot_SAP_000.pdf